CLINICAL TRIAL: NCT02087215
Title: Prospective Randomized Study of Local Application of Boron on Diabetic Foot Ulcers: Effect of Healing Process
Brief Title: Effect of Local Application of Boron on Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Mustafa Hasbahceci, surgeon, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRDIAFOOTULCER
Record Dates: First submitted 2014-01-28; First posted 2014-03-14 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetes mellitus; foot ulcer; boron; wound care
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer | interventions — Borates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- boron gel (Active Comparator): diabetic foot ulcer care with formulation gel: addition of borate as sodium penta boric acid pentahydrate 3% (w/v) and two different copolymer as pluronic block namely F68 2% (w/v) and f127 2% (w/v).
  Interventions: Drug: boron gel
- control gel (Placebo Comparator): placebo gel containing polymer of carbopol ultrex (1%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: boron gel — application of a formulation gel: addition of borate as sodium penta boric acid pentahydrate 3% (w/v) and two different copolymer as pluronic block namely F68 2% (w/v) and f127 2% (w/v) to diabetic foot ulcers.
  Other Names: borate as sodium penta boric acid pentahydrate 3%
  Arms: boron gel
Drug: Placebo
  Arms: control gel

SUMMARY:
Boron as a naturally occurring element has some metabolic and inflammatory actions. The antibacterial activity against gram negative bacteria is also known. Boron deficiency is shown to be related with impaired wound bone healing in rats. Therefore, special wound care formulas containing boron may have some positive effect on wound healing of the patients with diabetic foot ulcers.

DETAILED DESCRIPTION:
Local treatment of diabetic foot ulcers:

1. Classification of International Working Group of the Diabetic Foot (IWGDF)
2. pre-treatment measurements including diameter and area
3. pre-treatment laboratory values including fasting glucose, hemoglobin, hemoglobin A1c, leucocyte count and c-reactive protein
4. pre-treatment wound culture
5. treatment either by placebo gel containing polymer of carbopol ultrex (1%) or by formulation gel: addition of borate as sodium penta boric acid pentahydrate 3% (w/v) and two different copolymer as pluronic block namely F68 2% (w/v) and f127 2% (w/v).
6. post-treatment measurements and values

ELIGIBILITY:
Inclusion Criteria:

* diabetic food ulcer classified byInternational Working Group of the Diabetic Foot (IWGDF) as grade 1 and 2

Exclusion Criteria:

* previous vascular surgery on the side that the ulcer is present
* uncontrolled diabetes mellitus
* presence of osteitis, abscess, osteomyelitis, gangrene on the side that the ulcer is present
* diabetic food ulcer classified byInternational Working Group of the Diabetic Foot (IWGDF) as grade 3

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
number of the participants with complete epithelization of diabetic foot ulcer | up to 4 weeks
  healing and complete epithelization of diabetic foot ulcer with regard to time in weeks; comparison with progression or regression of grades of the wound based on classification sytems of International Working Group of the Diabetic Foot (IWGDF) and area of the wound measured as square centimeter.

SECONDARY OUTCOMES:
number of participants in whom local infective complications develop in diabetic foot ulcer patients | up to 4 weeks
  development of local infective complications including osteitis, abscess, osteomyelitis and gangrene

OTHER OUTCOMES:
improvement of inflammatory parameters in diabetic foot ulcers | up to 4 weeks
  improvement of inflammatory parameters in diabetic foot ulcers including leukocyte count, c-reactive protein and wound culture

CONTACTS AND LOCATIONS:
Overall Officials: mustafa hasbahceci, md, Principal Investigator — bezmialem vakif university faculty of medicine dept of general surgery
Locations (1):
- Mustafa Hasbahceci, Istanbul, Turkey (Türkiye)